CLINICAL TRIAL: NCT02585297
Title: The Presence of Microbes in the Sperm and Their Impact on Sperm Capacitation and IVF Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Meir hospital
Record Dates: First submitted 2015-10-08; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Semen and vaginal discharge
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Control- semen: Semen of fertile men
  Interventions: Other: no intervention
- Control- vaginal discharge: Vaginal discharge of partners of fertile men
  Interventions: Other: no intervention
- Case-semen: Semen of infertile men
  Interventions: Other: no intervention
- Case- vaginal discharge: Vaginal discharge of partners of infertile men
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Study Goals:

1. Finding the prevalence of bacteria of the sperm in an innovative and more accurate methode
2. Understanding the effect of microbes on the process of capacitation
3. The impact of microbes in the sperm on IVF success rate
4. Finding the incidence of vaginal bacteria and their relationship to bacteria of the sperm
5. The impact of vaginal flora on IVF success rate

DETAILED DESCRIPTION:
Prospective non interventional study in the Department of Life Sciences, Bar-Ilan University and IVF Unit at Meir Hospital.

The control group consisting of 50 semen samples from men with no sperm problems and 50 vaginal samples from their partners.

The study group consisting of 50 semen samples from men with male fertility problems and 50 vaginal samples from their partners.

The semen taken from the remains after fertilization of the IVF laboratory. (Liquid otherwise routinely thrown).

Vaginal samples taken from women undergoing IVF treatment under anesthesia after informed consent.

Enrollment also collect the following data: age, race, chronic illnesses, past surgeries and former fertility treatments. Data will be collected through anamnesis of the patient or the medical file after consent.

ELIGIBILITY:
Inclusion Criteria:

* Male and female undergoing fertility treatments

Exclusion Criteria:

* Male and female not undergoing fertility treatments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Infertile coupls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The percent of successful IFV treatments | 24 months
  Using 16-S Ribosomal RNA analysis to quantify and compare (type and percentages) of bacterial components in sperm samples from fertile and infertile men and their impact on IVF treatments success rate

REFERENCES:
- [Background] Trussell JC. Optimal diagnosis and medical treatment of male infertility. Semin Reprod Med. 2013 Jul;31(4):235-6. doi: 10.1055/s-0033-1345269. Epub 2013 Jun 17. No abstract available. PMID 23775377
- [Background] Rittenberg V, El-Toukhy T. Medical treatment of male infertility. Hum Fertil (Camb). 2010 Dec;13(4):208-16. doi: 10.3109/14647273.2010.534833. PMID 21117930
- [Background] Diemer T, Huwe P, Ludwig M, Hauck EW, Weidner W. Urogenital infection and sperm motility. Andrologia. 2003 Oct;35(5):283-7. PMID 14535856
- [Background] Goldenberger D, Kunzli A, Vogt P, Zbinden R, Altwegg M. Molecular diagnosis of bacterial endocarditis by broad-range PCR amplification and direct sequencing. J Clin Microbiol. 1997 Nov;35(11):2733-9. doi: 10.1128/jcm.35.11.2733-2739.1997. PMID 9350723
- [Background] Akutsu T, Motani H, Watanabe K, Iwase H, Sakurada K. Detection of bacterial 16S ribosomal RNA genes for forensic identification of vaginal fluid. Leg Med (Tokyo). 2012 May;14(3):160-2. doi: 10.1016/j.legalmed.2012.01.005. Epub 2012 Feb 7. PMID 22316585
- [Background] Domes T, Lo KC, Grober ED, Mullen JB, Mazzulli T, Jarvi K. The incidence and effect of bacteriospermia and elevated seminal leukocytes on semen parameters. Fertil Steril. 2012 May;97(5):1050-5. doi: 10.1016/j.fertnstert.2012.01.124. Epub 2012 Feb 16. PMID 22341372
- [Background] Bacteriospermia and sperm quality in infertile male patient
- [Background] De Francesco MA, Negrini R, Ravizzola G, Galli P, Manca N. Bacterial species present in the lower male genital tract: a five-year retrospective study. Eur J Contracept Reprod Health Care. 2011 Feb;16(1):47-53. doi: 10.3109/13625187.2010.533219. Epub 2010 Nov 23. PMID 21091298
- [Background] Hou D, Zhou X, Zhong X, Settles ML, Herring J, Wang L, Abdo Z, Forney LJ, Xu C. Microbiota of the seminal fluid from healthy and infertile men. Fertil Steril. 2013 Nov;100(5):1261-9. doi: 10.1016/j.fertnstert.2013.07.1991. Epub 2013 Aug 29. PMID 23993888
- [Background] Weng SL, Chiu CM, Lin FM, Huang WC, Liang C, Yang T, Yang TL, Liu CY, Wu WY, Chang YA, Chang TH, Huang HD. Bacterial communities in semen from men of infertile couples: metagenomic sequencing reveals relationships of seminal microbiota to semen quality. PLoS One. 2014 Oct 23;9(10):e110152. doi: 10.1371/journal.pone.0110152. eCollection 2014. PMID 25340531